CLINICAL TRIAL: NCT05573854
Title: Residual Gastric Volume After the Ingestion of an Oral Supplement Containing Carbohydrates and Whey Protein. A Randomized Crossover Pilot Study
Brief Title: Residual Gastric Volume After the Ingestion of Supplements Containing Carbohydrates and Whey Protein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Mato Grosso (Other)
Collaborators: Univag Centro Universitário (Other)
Responsible Party: Principal Investigator, José Eduardo de Aguilar-Nascimento, MD, PhD, Professor, Federal University of Mato Grosso
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 51807421.6.0000.5692
Record Dates: First submitted 2022-06-26; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Fasting; Gastric Stasis; Perioperative Complication; Safety Issues
Keywords: Preoperative care; Preoperative fasting; Whey protein; Gastric residual volume; Oral nutritional supplement
MeSH Terms: conditions — Fasting; Gastroparesis | interventions — Whey Proteins

STUDY DESIGN:
Intervention Model Description: The data will be collected in three phases. Firstly, after a fasting period of eight hours, the participants will attend the Radiology Service of the Hospital de Cancer, Cuiaba, Brazil to perform MRI images of the upper abdomen with the objective of measuring the fasting GRV (phase 1). In this phase, adequate stomach motility will be observed to exclude cases of possible gastroparesis. GRV (cmˆ3) will be measured in the fasting state by MRI tracking the region of interest (ROI) in each slice, forming a volume by the sum of all ROIs. In phase 2, each participant while still inside the MRI exam room will ingest 200 mL of the study drink described below. The individual will be immediately positioned in the supine position and another MRI scan will be carried out. Finally, phase 3 will be performed after a 3-hour pause and a third MRI scan will be done to measure again the GRV.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator will not participate of the 3 MRI sessions. Outcome Assessor will receive the data for statistical analysis blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Overnight Fast (Sham Comparator): After an overnight fast period of eight hours, the 6 participants will attend the Radiology Service of the Hospital de Câncer, Cuiaba, Brazil to perform MRI images of the upper abdomen with the objective of measuring the fasting GRV. GRV will be evaluated by tracking the region of interest (ROI) in each slice, forming a volume by the sum of all ROIs (phase 1).
  Interventions: Dietary Supplement: Overnight Fast
- Oral Supplement (Active Comparator): Each of the 6 participants while still inside the MRI exam room just after the MRI in fast condition, will ingest 200mL of the study oral supplement (OS). The individual will be immediately positioned in the supine position and another MRI scan will be carried out. In this second phase, GRV will be evaluated again as in phase 1 (phase 2).
  Interventions: Dietary Supplement: Gastric emptying after an oral supplement containing carbohydrates and whey protein
- 3h after ingestion (Active Comparator): Finally, phase 3 will be performed after a 3-hour pause. All volunteers, while still in the Radiology Service and fasted after the ingestion of the OS described in phase 2, will be submitted to a third MRI scan of the upper abdomen to measure again the GRV as previously described.
  Interventions: Dietary Supplement: Gastric emptying after an oral supplement containing carbohydrates and whey protein

INTERVENTIONS:
Dietary Supplement: Gastric emptying after an oral supplement containing carbohydrates and whey protein — Ingestion of an oral supplement containing carbohydrates and whey protein
  Arms: 3h after ingestion; Oral Supplement
Dietary Supplement: Overnight Fast — Residual Gastric Volume assessed by MRI after overnight fast (8h)
  Arms: Overnight Fast

SUMMARY:
Oral supplements (OS) containing carbohydrates are being used 2h before anesthesia. The addition of a nitrogen source would improve these drinks designed for the abbreviation of preoperative fasting. The gastric emptying of an oral supplement containing whey protein in addition to carbohydrates was investigated. This is a randomized crossover study including six healthy young volunteers who were submitted to abdominal MRI in 3 phases: 1) after a overnight fast, 2) after drank 200 mL of an OS containing whey protein and carbohydrates (no lipids), and 3) 3h after ingestion of the mentioned OS. The gastric residual volume (GRV) will be evaluate by MRI. The overall findings would allow us to conclude whether the GRV, assessed by MRI, in healthy young volunteers after three hours of the ingestion of 200 ml of an oral supplement containing carbohydrates associated with whey proteins is similar to the GRV found after an overnight fast. This pilot study will add important information to allow future randomized trials including an arm with patients undergoing elective surgical procedures with a 3h fasting after the ingestion of an OS containing whey protein and carbohydrates.

DETAILED DESCRIPTION:
One of most important prescription of enhanced recovery after surgery protocols is the reduction of preoperative fasting time in opposition to the traditional recommendation of overnight fast. This changing from prolonged fast to only 2-3h after the ingestion of 200-400 mL of carbohydrate (CHO)-enriched drinks in not only safe but recommended by various societies of anesthesia and nutrition. A long list of beneficial effects associated with the abbreviation of the preoperative fasting time with CHO beverages is reported ranging from alleviation of thirst, hunger and stress of the patient to metabolic benefits such as the improvement of insulin resistance. However, new formulas for preoperative beverages continue to evolve during the last years aiming to achieve better results. The addition of glutamine, anti-oxidants e recently whey protein to CHO-enriched formula has been tested and associated with a better reduction of insulin resistance, decrease of acute phase inflammatory response, and increasing production of glutathione. The effect of whey protein-enriched preoperative drinks on the postoperative functional capacity of patients are awaited. Nevertheless, only a few studies have tested the gastric emptying of drinks containing whey protein in addition to CHO Thus, the aim of this study is to investigate in healthy volunteers the gastric residual volume (GRV) 3h after ingesting a formula containing CHO and whey protein.

Methods This is an experimental pilot crossover clinical trial design.The data will be collected in three phases. Firstly, after a fasting period of eight hours, the participants attended the Radiology Service of the Hospital de Cancer, Cuiaba, Brazil to perform MRI images of the upper abdomen with the objective of measuring the fasting GRV (phase 1). In this phase, adequate stomach motility will be observed to exclude cases of possible gastroparesis that could interfere with gastric emptying and expected results. GRV (cmˆ3) will be measured in the fasting state as explained below. In phase 2, each participant while still inside the MRI exam room will ingest 200mL of the study drink described below. The individual will be immediately positioned in the supine position and another MRI scan will be carried out. In this second phase, GRV will be evaluated by tracking the same region of interest (ROI) in each slice, forming a volume by the sum of all ROIs. Finally, in phase 3 a third MRI scan of the upper abdomen to measure again the GRV as previously described will be done after a 3-hour pause.

Intervention oral supplement The oral supplement used as intervention for the study will be Nutren Fresh (Nestle, São Paulo, Brazil). This oral non-residual supplement (clear fluid) has 100% whey protein isolated from total proteins, with various vitamins (B1, B6, C, D, niacin and folic acid) with "lemon tea" flavor. In addition, the formula contains no lactose or lipids; is formulated with a volume of 200ml, with a caloric density of 1.28kcal/ml; protein: 10g in 200ml of product (100% whey protein isolate); and carbohydrate: 54g in 200ml of product (74% glucose syrup and 26% maltodextrin).

MRI Protocol All exams will be performed using the same MRI equipment which was a Magnetom Essenza 1.5T device; Siemens Healthcare, Brazil. Each volunteer will be placed in a supine position, with a body coil (Body Matrix) to capture the signal. Cross-sectional acquisitions with 40 slices (perpendicular to the longitudinal axis of the body) were performed in HASTE (echo-planar fast spin echo) sequences with a slice width of 4.0 mm at 3.0 mm intervals. This STEM sequence (TR [repetition time] 774 msec, TE [echo time] 92 msec) visualizes fluids with hypersignal as opposed to low signal from adjacent organs. Each acquisition of a set of images was performed during 15 seconds of apnea. The images will be captured by an industry technician with MRI experience and reviewed by a radiologist to confirm that the images covered the entire stomach. The GRV will be assessed by tracking the region of interest (ROI) in each slice, forming a volume by the sum of all ROIs. GRV measurements in cmˆ3 will be performed manually by tracing regions of interest on each slice using Osirix MD ANVISA v.12.0.3 software and summing the slices to determine total gastric volume and the results entered into an ExcelR data sheet for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Young
* Healthy volunteers

Exclusion Criteria:

* Gastroparesis
* Any gastrointestinal condition,
* Any chronic disease,
* Alcohol or any drug ingestion the day before of the MRI study
* Not completion of the 3 phases of the study protocol

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Gastric Residual Volume | 3 hours
  Gastric residual Volume in cmˆ3 assessed by MRI 3h after ingestion of the OS

CONTACTS AND LOCATIONS:
Overall Officials: Jose E Aguilar-Nascimento, MD, PhD, Principal Investigator — Univag Centro Universitário
Locations (1):
- Centro Universitário de Varzea Grande (UNIVAG), Várzea Grande, Mato Grosso, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Share will be possible by request via email
Supporting Information: Study Protocol, CSR
Time Frame: As soon as study is registered
Access Criteria: email

REFERENCES:
- [Background] de Aguilar-Nascimento JE, Caporossi C, Metelo JS, Tanajura GH, Canevari-de-Oliveira M, da Cunha Costa R. Safe intake of an oral supplement containing carbohydrates and whey protein shortly before sedation to gastroscopy; a double blind, randomized trial. Nutr Hosp. 2014 Mar 1;29(3):681-6. doi: 10.3305/nh.2014.29.3.7161. PMID 24559015
- [Background] Perrone F, da-Silva-Filho AC, Adorno IF, Anabuki NT, Leal FS, Colombo T, da Silva BD, Dock-Nascimento DB, Damiao A, de Aguilar-Nascimento JE. Effects of preoperative feeding with a whey protein plus carbohydrate drink on the acute phase response and insulin resistance. A randomized trial. Nutr J. 2011 Jun 13;10:66. doi: 10.1186/1475-2891-10-66. PMID 21668975
- [Background] Pimenta GP, de Aguilar-Nascimento JE. Prolonged preoperative fasting in elective surgical patients: why should we reduce it? Nutr Clin Pract. 2014 Feb;29(1):22-8. doi: 10.1177/0884533613514277. Epub 2013 Dec 11. PMID 24336400
- [Derived] Nogueira PLB, da Silva MR, Dock-Nascimento DB, de Aguilar-Nascimento JE. Residual gastric volume after 3 h of the ingestion of an oral supplement containing carbohydrates alone or associated with whey protein: a randomized crossover pilot study. Perioper Med (Lond). 2022 Dec 27;11(1):56. doi: 10.1186/s13741-022-00289-6. PMID 36575506